CLINICAL TRIAL: NCT03620786
Title: High-Intensity Focused Ultrasound for Focal Ablation of Prostate Tissue: An Observational Study of Multiparametric MRI and Ultrasound Fusion Imaging for Guidance
Brief Title: HIFU for Focal Ablation of Prostate Tissue: An Observational Study
Status: Recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Leonard S. Marks, M.D., Principal Investigator, University of California, Los Angeles
Other Study IDs: 16-000904
Record Dates: First submitted 2018-07-26; First posted 2018-08-08 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- HIFU Study Participants: Subjects who have biopsy-proven adenocarcinoma of the prostate, who have met all study inclusion and exclusion criteria, and have elected to receive or have already received the HIFU procedure as part of their routine prostate cancer treatment, will be invited to participate in this observational registry study. The HIFU device currently used in this standard-of-care procedure at UCLA is the Sonablate 450 HIFU System.
  Interventions: Device: Sonablate HIFU device

INTERVENTIONS:
Device: Sonablate HIFU device — In this study, we will be using the Sonablate 450 HIFU System. The Sonablate HIFU device was approved by the U.S. FDA for prostate tissue ablation in October, 2015. HIFU is an example of focal therapy, where the intervention involves targeting diseased areas of prostate tissue, while preserving healthy prostate tissue and minimizing damage to surrounding structures.

SUMMARY:
The Sonablate HIFU device was approved by the U.S.FDA for prostate tissue ablation in October, 2015. The purpose of this observational research study is to investigate the localized treatment of prostate cancer using HIFU through clinical data and health-related quality of life (HRQOL) questionnaires.

DETAILED DESCRIPTION:
This observational study will serve to collect data from medical record review and questionnaires before and after High Intensity Focused Ultrasound (HIFU) for focal ablation of prostate tissue. The subject will have already undergone or opted to receive the HIFU procedure as part of standard of care in order to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 years to 85 years
2. Subject has elected or already undergone HIFU therapy as their standard of care treatment methodand declined alternative treatment (active surveillance, radical prostatectomy, radiation therapy, cryosurgery and hormone therapy)
3. PSA ≤ 20
4. Prostate volume of ≤ 70 cc
5. Ability to complete informed consent form

Exclusion Criteria:

1. Prior treatment for prostate cancer (with the exception of androgen deprivation therapy)
2. Medical contraindication to follow-up mpMRI or prostate biopsy
3. Unable to tolerate general or regional anesthesia
4. Positive bone scan (only if bone scan has been done or clinically indicated. Bone scan does not need to be performed for study eligibility determination.)

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have biopsy-proven adenocarcinoma of the prostate, who have met all study inclusion and exclusion criteria, and have elected to receive or have already received the HIFU procedure as part of their routine prostate cancer treatment, will be invited to participate in this observational registry study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-26 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Oncological Response | 6 months
  The following definitions will be used for evaluation of oncological response:
  1. Complete response: Ablation of prostate tissue in targeted biopsy cores at 6 months and 18 months post-procedure biopsy and resolution of initial mp-MRI abnormality.
  2. Incomplete radiographic response: Residual mp-MRI abnormality at 6 months compared to baseline
  3. Local failure: Failure to ablate prostate tissue

SECONDARY OUTCOMES:
Evaluation of Quality-of-Life Symptoms (EPIC-CP) | 6 months
  The EPIC-CP questionnaire will be used to evaluate urinary, bowel and sexual health quality-of-life symptoms for participants pre- and post-HIFU.
Evaluation of Quality-of-Life Symptoms (EPIC-CP) | 18 months
  The EPIC-CP questionnaire will be used to evaluate urinary, bowel and sexual health quality-of-life symptoms for participants pre- and post-HIFU.
Decisional Regret Scale | 18 months
  This questionnaire data will be collected to assess for subjects' decision-making satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Marks, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No